CLINICAL TRIAL: NCT01678885
Title: Assessment of Energy Balance
Acronym: EnergyBalanc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 27007
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-02

CONDITIONS: Caloric Intake and Energy Metabolism
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sub-study 1, Dig Photo, Actical & IDEEA (Experimental): During one week of the doubly labeled water (DLW), participants will use digital photography of foods. During the other week of the DLW phase, participants will wear the Intelligent Device for Energy Expenditure and Activity (IDEEA) monitor and Actical monitor. Whether the participants wear the monitors first or complete digital photography first will be randomozed. Participants who complete the first two weeks and have a BMI over 25kg/m2 will receive a partial supplement low-calorie diet (LCD) for 8 weeks. This diet plan is a 1000-1150 kcal/day diet that participants will complete in a free-living environment. All participants will return to follow-up at six and twelve months after they completed the LCD. Anthropometric and questionnaire data will be collected.
  Interventions: Behavioral: Digital Photography of Foods; Other: doubly labeled water; Device: IDEEA; Behavioral: low-calorie diet; Device: Actical
- Sub-study 2 - Dig Photo & Sensewear (Experimental): During one week of the doubly labeled water (DLW) period, participants will use digital photography of foods. During the other week of the DLW phase, participants will wear the Sensewear armband. Whether the participants wear the monitor first or complete digital photography first will be randomozed. Participants who complete the first two weeks and have a BMI over 25kg/m2 will receive a partial supplement low-calorie diet (LCD) for 8 weeks. This diet plan is a 1000-1150 kcal/day diet that participants will complete in a free-living environment. All participants will return to follow-up at six and twelve months after they completed the LCD. Anthropometric and questionnaire data will be collected.
  Interventions: Behavioral: Digital Photography of Foods; Other: doubly labeled water; Behavioral: low-calorie diet; Device: Sensewear Armband

INTERVENTIONS:
Behavioral: Digital Photography of Foods — The digital photography of foods method was developed to unobtrusively measure energy intake in naturalistic settings (e.g., cafeterias). Participants will be provided with cell-phones with digital cameras and cellular network capability. Participants were trained to take pictures of their food selection and plate waste and to send these pictures to the researchers over the cellular network. The participant will collect data in free-living conditions and these data will be collected in near real time.
  Other Names: digital photography
Other: doubly labeled water — Doubly labeled water, considered the gold standard for measuring energy intake in humans, was used to measure total daily energy expenditure during free-living conditions. DLW is used to obtain an accurate measure of total daily energy expenditure, which is equal to energy intake during energy balance.
  Other Names: Doubly labeled water (DLW)
Device: IDEEA — The Intelligent Device for Energy Expenditure and Activity (IDEEA) will be used to measure the time spent engaging in active vs. sedentary behaviors, and the energy costs of these behaviors.
  Other Names: Intelligent Device for Energy Expenditure and Activity
  Arms: Sub-study 1, Dig Photo, Actical & IDEEA
Behavioral: low-calorie diet — Participants will be instructed to consume five packets of Health One per day, which provides 800 kcal and 125% of Recommended Daily Intake of vitamins and minerals. Additionally participants will be instructed to consume a meal consisting of 200 kcal to 350 kcal daily, which could consist of a portion-controlled meal replacement or a home-cooked meal. Participants will meet with a Registered Dietitian at weeks 0, 2, 4, and 6 and receive instructions on adhering to the meal plan.
  Other Names: LCD
Device: Actical — The Actical will be used to measure the time spent engaging in active vs. sedentary behaviors, and the energy costs of these behaviors.
  Arms: Sub-study 1, Dig Photo, Actical & IDEEA
Device: Sensewear Armband — The Sensewear armband will be used to measure the time spent engaging in active vs. sedentary behaviors, and the energy costs of these behaviors.
  Arms: Sub-study 2 - Dig Photo & Sensewear

SUMMARY:
The primary purpose of this study is to test different methods of measuring energy balance, including food intake and energy expenditure. Another primary purpose of this study is to see if energy expenditure predicts weight and change after a weight loss diet. A secondary aim will be to test the reliability and validity of the Actical accelerometer, SenseWear Armbands, and the Intelligent Device for Energy Expenditure and Activity (IDEAA) monitors at measuring activity energy expenditure (AEE) and total daily energy expenditure (TEE) against the gold standard, doubly-labeled water (DLW). Similarly, we will test whether the estimated energy expenditure or posture allocation from the 3 devices is associated with weight change during and following a low calorie diet (LCD).

DETAILED DESCRIPTION:
The study will take place over a period of one year. Participants will spend 3 weeks completing Phase I, and eight weeks completing Phase II (the weight loss phase of the study). Then, participants will return to the center at months 6 and 12 for a follow-up visit. During these visits, body weight, blood pressure, and pulse will be recorded, and questionnaires about eating attitudes and habits will be collected and assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Body Mass Index 25-40
* Willing to eat foods provided for two days.
* Willing to wear the IDEEA( Intelligent Device for Energy Expenditure and Activity), which is a device that attaches to the body and records movement and activity.
* Willing to wear an accelerometer, which is similar to a pager that attaches to belt or clothing and measures activity.
* Willing to use a cell phone equipped with a digital camera to take pictures of foods for one week.
* Willing to undergo an 8 week weight loss diet, consisting of supplement or powdered shakes, portion-controlled entrees, or home-cooked meals.

Exclusion Criteria:

* A diagnosis of diabetes, cardiovascular disease, or cancer.
* Females who are pregnant or planning to become pregnant during the trail.
* Medications that influence appetite or body weight (weight loss medications such as sibutramine, antipsychotic medications such as olanzapine, or herbal weight loss products) taken during the previous three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corby K Martin, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Sub-study 1 - Dig Photo First, Then IDEEA & Actical; Phase 1 Sub-study 1 - IDEEA & Actical First, Then Dig Photo; Phase 1 Sub Study 2 - Dig Photo First, Then Sensewear: Participants completed 2 phases of the study. Phase I included a 2-week doubly labeled water period where they also wore activity trackers for one week, and used a food photography method for the other week. Phase II was an 8-week partial supplement low-calorie diet (LCD). This diet plan was a 1000-1150 kcal/day diet composed of HealthOne shakes and prepackaged portion controlled foods or home-cooked meals that participants completed in a free-living environment. Participants returned to follow-up at six and twelve months after they completed the LCD. During these assessments, anthropometric and questionnaire data were collected.
- Phase I Sub Study 2 - Sensewear First, Then Digital Photo: Phase 1- sensewear First, Then Digital Photography
- Phase 2- Low-Calorie Diet: Participants from sub-study 1 and 2 had the chance to receive the low-calorie diet based on their eligibility; i.e., BMI level.
  Participants completed 2 phases of the study. Phase I included a 2-week doubly labeled water period where they also wore activity trackers for one week, and used a food photography method for the other week. Phase II was an 8-week partial supplement low-calorie diet (LCD). This diet plan was a 1000-1150 kcal/day diet composed of HealthOne shakes and prepackaged portion controlled foods or home-cooked meals that participants completed in a free-living environment. Participants returned to follow-up at six and twelve months after they completed the LCD. During these assessments, anthropometric and questionnaire data were collected.
Period: Phase I; 2 Wks Duration, Both Sub-study
Arm/Group | Phase I Sub-study 1 - Dig Photo First, Then IDEEA & Actical | Phase 1 Sub-study 1 - IDEEA & Actical First, Then Dig Photo | Phase 1 Sub Study 2 - Dig Photo First, Then Sensewear | Phase I Sub Study 2 - Sensewear First, Then Digital Photo | Phase 2- Low-Calorie Diet
Started | 22 | 18 | 23 | 24 | 0
Completed | 22 | 15 | 22 | 21 | 0
Not Completed | 0 | 3 | 1 | 3 | 0
Period: Phase II; 8 Week Low Calorie Diet
Arm/Group | Phase I Sub-study 1 - Dig Photo First, Then IDEEA & Actical | Phase 1 Sub-study 1 - IDEEA & Actical First, Then Dig Photo | Phase 1 Sub Study 2 - Dig Photo First, Then Sensewear | Phase I Sub Study 2 - Sensewear First, Then Digital Photo | Phase 2- Low-Calorie Diet
Started | 0 | 0 | 0 | 0 | 87
Completed | 0 | 0 | 0 | 0 | 70
Not Completed | 0 | 0 | 0 | 0 | 17

BASELINE CHARACTERISTICS:
Groups:
- Sub-study 1; Sub-study 2: During the first week of the doubly labeled water period (day 0 to 7), participants in group 1 will use digital photography of foods. During the second week of the doubly labeled water phase, participants in this group will wear the Intelligent Device for Energy Expenditure and Activity (IDEEA) monitor and an accelerometer.During the first week of the doubly labeled water period (day 0 to 7),participants in group 2 will wear the IDEEA monitor and accelerometer in the first week of the doubly labeled water period and digital photography of foods during the second week.Participants who complete Phase I of the study will receive a partial supplement low-calorie diet (LCD) for 8 weeks. Participants will return to follow-up at six and twelve months after they completed the LCD. During these assessments, anthropometric and questionnaire data will be collected.
- Total: Total of all reporting groups
Arm/Group | Sub-study 1 | Sub-study 2 | Total
Number analyzed (Participants) | 40 | 47 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 47 | 87
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 41 | 72
  Male | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 40 | 47 | 87

OUTCOME MEASURES:

1. Primary Outcome: ENERGY BALANCE EQUATION, PHASE I, ONE SUB-STUDY
Description: A new method of digital photography of foods to measure the energy intake (EI) and macronutrient intake of free-living humans was tested. Digital photography (RFPM) EI was tested against measured food provisions during an in-feeding period and against EI measured with doubly labeled water (DLW) during free-living conditions for 1 week. EI measured by directly weighing food provisions in the clinic over two days and measuring food intake during free-living conditions over one week with the DLW.
Time Frame: ~6 days
Population: Free-living energy intake data were analyzed from the 40 participants who completed the protocol and provided urine samples for doubly labeled water analysis. This primary outcome measure was limited to one sub-study.
Measure: Mean (Standard Deviation); unit: kCal
Groups:
- Phase 1: During the first week of the doubly labeled water period (day 0 to 7), participants in group 1 will use digital photography of foods (RFPM). During the second week of the doubly labeled water phase, participants in this group will wear the Intelligent Device for Energy Expenditure and Activity (IDEEA) monitor and an accelerometer. Participants in group 2 will wear the IDEEA monitor and accelerometer in the first week of the doubly labeled water period and digital photography of foods during the second week.
Arm/Group | Phase 1
Number analyzed (Participants) | 42
kCal
  EI (kcal) Measured with DLW | 2360 (626)
  EI (kcal) Measured with RFPM | 2208 (665)
  Difference of EI (kcal) measured with DLW and RFPM | -152 (694)

2. Secondary Outcome: Weight Change
Description: The secondary aim was to test if posture allocation (the amount of time spent engaging in certain behaviors e.g., sitting, walking, running, changing positions and the energy burned during these activities) predicts weight change over one year following a period of weight loss.
Time Frame: 1 year
Population: Weight change was evaluated from all participants who received the low calorie diet in sub-studies 1 and 2 combined.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Phase II: Participants who complete Phase I of the study received a partial supplement low-calorie diet (LCD) for 8 weeks. This diet plan was a 1000-1150 kcal/day diet composed of Health One shakes and prepackaged portion controlled foods or home-cooked meals that participants completed in a free-living environment. Participants returned to follow-up at six and twelve months after they completed the LCD. During these assessments, anthropometric and questionnaire data was collected.
Arm/Group | Phase II
Number analyzed (Participants) | 53
kg | -6.3 (2.1)

3. Secondary Outcome: Total Energy Expenditure (TEE) and Activity Energy Expenditure (AEE) Predictions From Actical, IDEEA, and Sensewear Monitors (kcal/Day)
Description: Bland-Altman analyses compared the TDEE and AEE from the Sensewear® and IDEEA and Actical monitors to the DLW data from the week participants wore the monitors. Only the week of DLW data that corresponded with the wearing of the monitors was used for this analysis.
Time Frame: 1 week
Population: Of the 87 participants considered from phase 1 of sub-studies 1 and 2, five were excluded because they did not finish baseline accelerometry assessment, five were excluded because they did not enter the LCD due to BMI's < 25. Seven were excluded because they did not successfully complete all aspects of the DLW dosing period.
Measure: Mean (Standard Deviation); unit: kcal/day
Groups:
- All Participants: During the first week of the doubly labeled water period (day 0 to 7), participants in group 1 will use digital photography of foods. During the second week of the doubly labeled water phase, participants in this group will wear the Intelligent Device for Energy Expenditure and Activity (IDEEA) monitor and an accelerometer.During the first week of the doubly labeled water period (day 0 to 7),participants in group 2 will wear the IDEEA monitor and accelerometer in the first week of the doubly labeled water period and digital photography of foods during the second week.Participants who complete Phase I of the study will receive a partial supplement low-calorie diet (LCD) for 8 weeks. Participants will return to follow-up at six and twelve months after they completed the LCD. During these assessments, anthropometric and questionnaire data will be collected.
Arm/Group | All Participants
Number analyzed (Participants) | 70
kcal/day
  kcal/day; Sensewear TEE | -59.98 (411.5)
  kcal/day, IDEEA TEE | 121.72 (467.8)
  kcal/day, Actical Waist AEE | -111.38 (354.1)
  kcal/day, Actical Wrist AEE | 194.52 (454.0)
  kcal/day, Sensewear AEE | -416.95 (370.6)
  kcal/day, IDEEA AEE | 108.77 (436.8)

4. Secondary Outcome: Device Predictions of % Weight Change During and After an 8-week LCD
Description: This secondary aim of the study was evaluated with linear regression analysis to determine if TEE, AEE, or measures of posture allocation predicted weight loss during the 8-week LCD. Percent weight change from diet initiation to termination was the dependent variable for the weight loss regressions. Of the 87 participants considered for these secondary analyses, five were excluded because they did not finish baseline accelerometry assessment, and an additional five were excluded because they did not enter the LCD phase due to BMI's < 25. Finally, seven more participants from this original sample were excluded because they did not successfully complete all aspects of the DLW dosing period. Finally, an additional 4 subjects were lost to follow up during the 8-week LCD period. Thus, 66 participants were included in the analysis
Time Frame: 8 weeks
Population: Participants from sub-study 1 and 2 combined were used in this analysis.
Measure: Number; unit: R squared
Groups:
- All Participants: All study participants were included in these analyses
Arm/Group | All Participants
Number analyzed (Participants) | 66
R squared
  Actical (waist) AEE | 0.00
  Actical (wrist) AEE | 0.00
  Sensewear TEE | 0.00
  Sensewear AEE | 0.10
  IDEEA TEE | .03

ADVERSE EVENTS:
Description: Adverse events reported for Phase 1 and 2. Participants are stratified by the sub-studies.
Groups:
- Sub-study 1; Sub-study 2: Participants completed 2 phases of the study. Phase I included a 2-week doubly labeled water period where they also wore activity trackers for one week, and used a food photography method for the other week. Phase II was an 8-week partial supplement low-calorie diet (LCD). This diet plan was a 1000-1150 kcal/day diet composed of HealthOne shakes and prepackaged portion controlled foods or home-cooked meals that participants completed in a free-living environment. Participants returned to follow-up at six and twelve months after they completed the LCD. During these assessments, anthropometric and questionnaire data were collected.
Arm/Group | Sub-study 1 | Sub-study 2
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/47
Other Adverse Events (participants affected / at risk) | 0/40 | 0/47

LIMITATIONS AND CAVEATS:
The study included a 2-week doubly labeled water phase; hence, the activity and energy intake assessments were limited this period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No